CLINICAL TRIAL: NCT04714996
Title: A Phase 2A, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Pharmacokinetics of ES-481 in Adult Patients With Drug Resistant Epilepsy
Brief Title: Efficacy, Safety and Pharmacokinetics of ES-481 in Adult Patients With Drug Resistant Epilepsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ES Therapeutics Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ES-481-C201
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ES-481 (Experimental)
  Interventions: Drug: ES-481
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Open-Label Extension Study (Other)
  Interventions: Drug: Open-Label Extension Study

INTERVENTIONS:
Drug: ES-481 — Treatment Period Week 1 - 25 mg qd, Week 2 - 25 mg bid, Week 3 - 50 mg bid, Week 4 - 75 mg bid.
  Step-down and Washout Period Day 1 - 125 mg, Day 2 - 100 mg, Day 3 - 75 mg, Day 4 - 50 mg, Day 5 - 50 mg, Day 6 - 25 mg, Day 7 - 25 mg, Days 8 to 14 - 0 mg
  Arms: ES-481
Drug: Placebo — Placebo on Week 1, Week 2, Week 3 and Week 4
  Arms: Placebo
Drug: Open-Label Extension Study — Dosing will be at the discretion of the Investigator with a minimum dose of 25 mg/day (25 mg qd) to a maximum dose of 150 mg/day (75 mg bid).
  Arms: Open-Label Extension Study

SUMMARY:
This is a Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study with cross-over to Evaluate the Efficacy, Safety, and Pharmacokinetics of ES-481 in Adult Patients with Drug Resistant Epilepsy

ELIGIBILITY:
Inclusion Criteria:

1. The subject/legal guardian must be able to understand and sign the Human Research Ethics Committee-approved written Informed Consent Form (ICF) and privacy language as per national regulations (e.g., HREC and TGA requirement in Australia) prior to any study-related procedures being performed
2. The subject is a male or female 18 to 70 years of age, inclusive
3. The subject must have a history of drug resistant epilepsy (as per the ILAE definition)
4. The subject must be taking 1 to 4 antiepileptic drugs (AED) and must be on a stable dose of the AEDs for at least four (4) weeks prior to entering the 28-day screening period
5. If VNS implanted, the stimulation setting must have been stable for at least four weeks prior to entering the 28-day screening period
6. The subject/legal guardian must be able to use the seizure dairy to record seizure throughout the study
7. The subject must experience at least four (4) countable seizures within a 28-day period.

   For continued enrollment into Treatment Period 1, each subject will be confirmed to have experienced at least four (4) countable seizures in the 28-day screening period
8. The subject must have interictal epileptiform discharges and/or seizure with an average frequency of at least one (1) per hour on EEG recording.

   For continued enrollment into Treatment Period 1, this will be confirmed by a 24-hour EEG performed during the 28-day screening period.
9. The subject is willing and able to comply with the study requirements

Exclusion Criteria:

1. Unwilling or inability to follow the procedures specified by the protocol
2. Pregnancy or breast feeding
3. Women of child-bearing potential and men who are unable or unwilling to take adequate contraceptive precautions, including one of the following:

   Hormonal contraception (birth control pills, injected hormones or vaginal ring) Intrauterine device Barrier methods (condom or diaphragm) combined with spermicideSurgical sterilization (hysterectomy, tubal ligation, or vasectomy)
4. Current treatment for another significant medical disorder, such as diabetes, or heart disease or an untreated disorder, that is discovered during the 28-day screening period and might interfere with the study in the opinion of the Principal Investigator
5. An abnormality on clinical laboratory tests, physical examination, EEG or ECG that might increase the risks associated with trial participation or investigational product administration, such as hepatic enzyme elevation greater than twice normal and/or a GFR < 60 mL/min/1.73 m2
6. History (within the month) of illicit drug use or alcohol dependence, and a commitment by the subject to not take the illicit drugs during the study
7. Concomitant treatment with more than four (4) AEDs
8. Evidence for a potentially progressive neurologic disorder, such as a brain tumor, multiple sclerosis or dementia
9. Planned epilepsy surgery within six months of enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Seizure Frequency | Continuous and at Days 1, 8, 15, 22, 28, 43, 50, 57, 64 and 70
  A change in seizure frequency and activity assessed using a patient diary and continuous 24-hour EEG monitoring (composite outcome)

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | Collected at screening, Days 1, 8, 15, 22, 28, 43, 50, 57, 64 and 70
  To assess for changes in the HAM-A
Hamilton Depression Rating Scale (HDRS) | Collected at screening, Days 1, 8, 15, 22, 28, 43, 50, 57, 64 and 70
  To assess for changes in HDRS
Adverse Events | Collected at screening, Days 1, 8, 15 22, 28, 43, 50, 57, 64 and 70
  Monitoring clinically for adverse events for both CNS and Cardiovascular events
Laboratory Assessments - Hematology | Collected at screening, Days 1, 8, 15 22, 28, 43, 50, 57, 64 and 70
  Assess changes in hematology and chemistry laboratories by blood and serum assays and analysis
Laboratory Assessments - Chemistry | Collected at screening, Days 1, 8, 15 22, 28, 43, 50, 57, 64 and 70
  Assess changes in hematology and chemistry laboratories by blood and serum assays and analysis
Pharmacokinetics (PK) - Cmax | Collected at screening, Days 1, 8, 15 22, 28, 43, 50, 57, 64 and 70
  Plasma concentration-time data will be analyzed using non compartmental methods to determine the following PK parameter: Cmax
Pharmacokinetics (PK) - Tmax | Collected at screening, Days 1, 8, 15 22, 28, 43, 50, 57, 64 and 70
  Plasma concentration-time data will be analyzed using non compartmental methods to determine the following PK parameter: Tmax
Pharmacokinetics (PK) - AUC0-t | Collected at screening, Days 1, 8, 15 22, 28, 43, 50, 57, 64 and 70
  Plasma concentration-time data will be analyzed using non compartmental methods to determine the following PK parameter: AUC0-t
Pharmacokinetics (PK) - AUC0-inf. T1/2 | Collected at screening, Days 1, 8, 15 22, 28, 43, 50, 57, 64 and 70
  Plasma concentration-time data will be analyzed using non compartmental methods to determine the following PK parameter: AUC0-inf. T1/2
Pharmacokinetics (PK) - CL/F | Collected at screening, Days 1, 8, 15 22, 28, 43, 50, 57, 64 and 70
  Plasma concentration-time data will be analyzed using non compartmental methods to determine the following PK parameter: CL/F
Pharmacokinetics (PK) - Vz/F | Collected at screening, Days 1, 8, 15 22, 28, 43, 50, 57, 64 and 70
  Plasma concentration-time data will be analyzed using non compartmental methods to determine the following PK parameter: Vz/F

CONTACTS AND LOCATIONS:
Overall Officials: Terence O'Brien, Principal Investigator — The Alfred
Locations (4):
- Australia (4):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria